CLINICAL TRIAL: NCT06719843
Title: Effectiveness of an Acceptance and Commitment Therapy-based Intervention in Reducing Loneliness Among Older Adults Living Alone: a Cluster-randomised Wait-list Controlled Trial
Brief Title: Acceptance and Commitment Therapy-based Intervention for Loneliness Among Older Adults Living Alone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Salvation Army, Hong Kong and Macau Command (Other)
Responsible Party: Principal Investigator, Cho Lee Wong, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024.026-T
Record Dates: First submitted 2024-11-27; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Loneliness
Keywords: Loneliness; Older adults; Acceptance and committment therapy-based intervention

STUDY DESIGN:
Intervention Model Description: Wait-list trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACT-based intervention (Experimental): In addition to usual community support services, participants in the intervention group will receive the face-to-face ACT-based intervention weekly for 4 weeks (each session lasting approximately 90 minutes), with each group consisting of 6-8 older adults.
  Interventions: Behavioral: ACT-based intervention
- Wait-list control (No Intervention): Participants in the wait-list control group will receive usual community support services (e.g. meal delivery) provided by the community centres they belong to.

INTERVENTIONS:
Behavioral: ACT-based intervention — Participants in the intervention group will receive the face-to-face ACT-based intervention weekly for 4 weeks (each session lasting approximately 90 minutes), with each group consisting of 6-8 older adults. The intervention consists of 4 sessions:
  Session 1 (acceptance and cognitive fusion) Session 2 (contact with the present moment and self-as-context) Session 3 (values) Session 3 (committed action)
  Arms: ACT-based intervention

SUMMARY:
The proposed cluster-randomised wait-list-controlled trial will (1) examine the effects of the acceptance and commitment therapy (ACT)-based intervention on loneliness, psychological flexibility, psychological distress, health-related quality of life, and healthcare utilisation among older adults living alone in Hong Kong; (2) investigate whether the effect of the ACT-based intervention on loneliness is mediated through psychological flexibility; and (3) explore the experiences and perceptions of older adults living alone who participate in ACT-based interventions, including their perceptions of the intervention's impact on their loneliness.

DETAILED DESCRIPTION:
A convenience sample of 234 older adults living alone will be recruited from six participating community centres (39 participants from each centre). Eligible older adults will be randomly assigned to a waitlist control group (n = 117) or an intervention group (n = 117). Both groups will receive usual community support services. The intervention group will additionally receive four weekly face-to-face ACT-based intervention sessions (approximately 90 minutes each) in group format (each group consisting of six to eight older adults).

The primary outcome (loneliness) and secondary outcomes (psychological flexibility, psychological distress, health-related quality of life, and healthcare utilisation) will be assessed at baseline (T0), immediately post-intervention (T1), 3 months post-intervention (T2) and 6 months post-intervention (T3), using validated questionnaires. A purposive subsample of 36 intervention group participants will be invited for focus group interviews. A generalised estimating equation model with intention-to-treat and path analyses will be used to analyse the quantitative data, whereas thematic analysis will be used for the qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* older adults aged 60 years or above
* residing in the community (living at home without being institutionalised in the past 6 months)
* capable of speaking and understanding Chinese
* experiencing loneliness (scoring ≥3 on a three-item loneliness screening scale)
* living alone for more than 1 year

Exclusion Criteria:

* currently undergoing psychological intervention
* having a clinical diagnosis of mental illness
* being cognitively impaired (Abbreviated Mental Test score <6)
* having visual/language/communication difficulties

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Loneliness | Assessed at baseline (T0), within 1 day (T1), 3 months (T2), and 6 months (T3) after the completion of the intervention
  The Chinese version of the six-item De Jong Gierveld Loneliness Scale (DJGLS) will be used to measure loneliness. This scale comprises six items measuring emotional and social loneliness. The scores range from 0 to 6, a higher score indicates a greater level of loneliness.

SECONDARY OUTCOMES:
Psychological flexibility | Assessed at baseline (T0), within 1 day (T1), 3 months (T2), and 6 months (T3) after the completion of intervention
  The short form of the Comprehensive assessment of Acceptance and Commitment Therapy Processes will be used to measure psychological flexibility. It comprises 10 items measuring openness to experience, behavioural awareness, and valued action. The scores range from 0 to 60. A higher score indicates greater psychological flexibility.
Psychological distress | Assessed at baseline (T0), within 1 day (T1), 3 months (T2), and 6 months (T3) after the completion of the intervention
  The Chinese version of the Depression Anxiety Stress Scale (DASS-21) will be used to measure psychological distress. It comprises 21 items measuring depressive, anxiety, and stress symptoms in older adults. A higher score indicates a higher level of psychological distress. The cutoff scores that indicate severe and highly severe depression, anxiety, and stress are >20, >14, and >25, respectively.
Health-related quality of life | Assessed at baseline (T0), within 1 day (T1), 3 months (T2), and 6 months (T3) after the completion of intervention
  The Chinese (Hong Kong) Short Form-12 version 2 (SF-12v2) will be used to assess health-related quality of life (HRQOL). It comprises 12 items that measure eight domains of quality of life, which are summed into two subscales. The scores range from 0 to 100. A high score indicates good HRQOL.
Healthcare utilisation | Assessed at baseline (T0), within 1 day (T1), 3 months (T2), and 6 months (T3) after the completion of intervention
  It will be assessed based on the number of accident and emergency department visits, outpatient clinic visits (e.g., specialist outpatient clinic, family medicine, general outpatient clinic, and allied health appointments), and inpatient length of stay.
Experiences and perceptions of older adults in intervention group | Assessed within 1 day (T1) after the intervention
  Focus group interviews will be conducted to explore the experiences and perceptions of older adults in intervention group regarding their participation in ACT-based interventions and the impact of the intervention on their loneliness using an interview guide.

IPD SHARING:
Plan to Share IPD: No